CLINICAL TRIAL: NCT05375461
Title: A Phase III,randomized, Double-blind, Paralle, Multi-center Study to Evaluate the Efficacy and Safety of TQB3616 Capsules Plus Fulvestrant Compared to Placebo Plus Fulvestrant in Participants with Hormone Receptor (HR)-positive, Human Epidermal Growth Factor Receptor(EGFR) 2-Negative Advanced Breast Cancer
Brief Title: TQB3616 Capsules Plus Fulvestrant Compared to Placebo Plus Fulvestrant in Previously Treated Breast Cancer in Clinical Trail
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB3616-III-01
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HR-positive,HER2-negative in Advanced Breast Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TQB3616 capsules plus fulvestrant (Experimental): The dose of TQB3616 capsules is 180mg, taken orally on an empty stomach, once a day for 28 consecutive days as one treatment cycle.
  Fluvestrin injection was given at a fixed dose of 500mg on day 1, day 15 of the first treatment cycle and day 1 of each subsequent treatment cycle, and a treatment cycle of 28 days.
  Interventions: Drug: TQB3616 capsules; Drug: Fluvestrin injection
- TQB3616-matching placebo plus fulvestrant (Placebo Comparator): The dose of placebo is 180mg, taken orally on an empty stomach, once a day for 28 consecutive days as one treatment cycle.
  Fluvestrin injection was given at a fixed dose of 500mg on day 1, day 15 of the first treatment cycle and day 1 of each subsequent treatment cycle, and a treatment cycle of 28 days.
  Interventions: Drug: TQB3616-matching placebo; Drug: Fluvestrin injection

INTERVENTIONS:
Drug: TQB3616 capsules — The dose of TQB3616 capsules is 180mg, taken orally on an empty stomach, once a day for 28 consecutive days as one treatment cycle.
  Arms: TQB3616 capsules plus fulvestrant
Drug: TQB3616-matching placebo — The dose of placebo is 180mg, taken orally on an empty stomach, once a day for 28 consecutive days as one treatment cycle.
  Arms: TQB3616-matching placebo plus fulvestrant
Drug: Fluvestrin injection — Fluvestrin injection was given at a fixed dose of 500mg on day 1, day 15 of the first treatment cycle and day 1 of each subsequent treatment cycle, and a treatment cycle of 28 days.

SUMMARY:
This is a Phase III, a randomized, double-blind, parallel , multi-center trail to evaluate the efficacy and safety of TQB3616 capsules plus fulvestrant compared to placebo plus fulvestrant in participants with estrogen receptor-positive, HER2-Negative Advanced Breast Cancer. Approximately 287 women will be randomized to either TQB3616 plus fulvestrant or TQB3616-matching placebo plus fulvestrant. Randomization will follow a 2:1 randomization ratio,the experimental is 191; the Placebo Comparator is 96.

ELIGIBILITY:
Inclusion Criteria:

* 1 The subjects voluntarily joined the study and signed the informed consent, with good compliance.
* 2 Age: 18-75 years old (upon signing the informed consent);ECOG PS score: 0~1; Expected survival ≥3 months.
* 3 participants with estrogen receptor-positive, HER2-Negative Advanced Breast Cancer were identified by pathological testing.
* 4 Patients at the relapse/metastatic stage were allowed to receive no more than 1 line of rescue chemotherapy or rescue endocrine therapy.
* 5 Confirmation of at least one measurable lesion according to RECIST1.1 criteria.
* 6 The main organs are functioning well and meet the following criteria: Routine blood examination criteria (no blood transfusion or hematopoietic stimulus drug correction within 7 days before screening) : a) hemoglobin (Hb) ≥100g/L; b) neutrophils absolute value (NEUT) ≥1.5×10^9/L; c) Platelet count (PLT) ≥90×10^9/L.

Biochemical tests should meet the following criteria: a) Total bilirubin (TBIL) ≤2.5 times the upper limit of normal (ULN); b) Alanine transferase (ALT) and aspartate transferase (AST) ≤2.5×ULN.ALT and AST≤5×ULN with liver metastasis. c) Serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance rate (CCR) ≥60ml/min.

The blood coagulation function test should meet the following criteria: prothrombin time (PT), activated partial thromboplastin time (APTT), international standardized ratio (INR) ≤1.5×ULN (no anticoagulant therapy); Cardiac ultrasound evaluation: left ventricular ejection fraction (LVEF)≥50%.

Exclusion Criteria:

* 1 Complicated diseases and medical history:

  1. Has had other malignant tumors within 3 years or currently has other malignant tumors;
  2. Have a variety of factors that affect oral medication (such as inability to swallow, chronic diarrhea, and intestinal obstruction);
  3. Unmitigated toxicity above CTCAE1 grade due to any prior treatment;
  4. Severe infections (≥CTCAE2 grade) that were active or uncontrolled before the study treatment started;
  5. Cirrhosis, active hepatitis；
  6. Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
* 2 Tumor-related symptoms and treatment:

  1. Clinical evidence or history of central nervous system metastases (CNS) and/or cancerous meningitis or pneumomeningeal disease;
  2. Had received chemotherapy within 3 weeks prior to the start of study treatment, and had received radiotherapy (except palliative radiotherapy for non-target lesions), hormone therapy, or other anti-tumor therapy within 2 weeks prior to the start of study treatment (washout period was calculated from the end of last treatment);
  3. Uncontrolled pleural effusion, pericardial effusion, or ascites that still require repeated drainage (as determined by the investigator).
* 3 Known to be allergic to fluvestone, TQB3616 or any excipient.
* 4 Participated in clinical trials of other antitumor drugs within 4 weeks prior to the initiation of study therapy.
* 5 Has other conditions that make it inappropriate for the patient to be enrolled based on investigator's opinion.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Baseline up to 24 months
  Progression-free survival (First-time progression of disease/ recurrence /death)

SECONDARY OUTCOMES:
Progression-free survival (PFS) by Independent Review Committee | Baseline up to 24 months
  Progression-free survival（First-time progression of disease/ recurrence /death）
Overall survival (OS) | Baseline up to 24 months
  Overall survival (Baseline up to death)
Clinical benefit rate (CBR) | Baseline up to 24 months
  Percentage of subjects with complete (CR) or partial response (PR) or stable disease (SD)（ Baseline up to progression of disease/ recurrence /death）
Duration of Response (DOR) | Baseline up to 24 months
  Duration of Response(Baseline up to progression of disease/ recurrence /death)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hosptital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yin Y, Zhang Q, Sun T, Hao C, Wang Z, Yang J, Wang Y, Shi Y, Sun J, Ouyang Q, Su H, Wu J, Gan L, Han M, Gao L, Wang X, Zhao B, Li H, Zhao J, Yang H, Ning F, Tian F, Zhang J, Sun H, Niu Z, Zong H, Zang A, Wang X, Qian X, Wu S, Nie J, He L, Cheng Y, Hao Y, Zhai Y, Li H, Wang J, Wei S, Li M, Liu Y, Guo H, Hu Q, Liu L, Han X, Luo R, Ni M, Tang X, Zhai Z, Ding M, Wang H, Shen P, Wang X, Liu L, Chen W, Liu G, Cai Z, Jiang Z. Novel CDK2/4/6 inhibitor culmerciclib (TQB3616) plus fulvestrant in previously treated, HR-positive, HER2-negative advanced breast cancer: a randomized, double-blind, phase 3 trial. Signal Transduct Target Ther. 2025 Dec 18;10(1):414. doi: 10.1038/s41392-025-02475-6. PMID 41413016
- [Derived] Xu Z, Liu Y, Song B, Ren B, Xu X, Lin R, Zhu X, Chen C, Yang S, Zhu Y, Jiang W, Li W, Xia Y, Hu L, Chen S, Chan CC, Li J, Zhang X, Yang L, Tian X, Ding CZ. Discovery and preclinical evaluations of TQB3616, a novel CDK4-biased inhibitor. Bioorg Med Chem Lett. 2024 Jul 15;107:129769. doi: 10.1016/j.bmcl.2024.129769. Epub 2024 Apr 24. PMID 38670537